CLINICAL TRIAL: NCT02619045
Title: Evaluation of the Impact of a Follow-up Phone Call Nurse Device in the Care of Patients With Chemotherapy Treatment, in Their Quality of Life and Medico-economic Analysis of This Follow-up Program Device
Brief Title: Evaluation of the Impact of a Follow-up Phone Call Nurse Device in the Care of Patients With Chemotherapy Treatment
Acronym: EVAL'COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14 GENE 07
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solid tumors (Other): Patients with solid tumor starting a intra venous chemotherapy with 21 days cycles.
  Interventions: Other: Telephone follow-up nursing device

INTERVENTIONS:
Other: Telephone follow-up nursing device — Telephone follow-up nursing device involving:
  * telephone appointments made by a dedicated nurse and set up at key stage of treatment (1 phone call per week during chemotherapy cycles),
  * specific questionnaire used by the nurse at each phone call (toxicity, general care, quality of life...),
  * actions taken for the patient following each phone call (consultation with a doctor, patient hospitalization, sending of a prescription, coordination with the city medical caregiver);

SUMMARY:
This study evaluate the Impact of a Follow-up Phone Call Nurse Device in the Care of Patients With Chemotherapy Treatment, in their Quality of Life and Medico-economic Analysis of this Follow-up Program Device.

DETAILED DESCRIPTION:
This study is a monocentric prospective cohort study designed to monitor the care of patients undergoing an intra venous chemotherapy. Patients with a solid tumor (200 patients in total), starting a first cycle of intravenous chemotherapy with 21 days cycle will be included in this study. Patients will be followed all over the chemotherapy period through regular and defined telephone appointments carried out by a dedicated nurse. During phone call, a specific questionnaire will be used in order to retrieve data regarding patients toxicities, general care, quality of life, ...Actions taken following each phone call will also be documented (consultation, hospitalization, prescription,...). The main objective of this study is to evaluate the impact of this telephone follow-up program on the care of patients under chemotherapy treatment. In addition, a medico-economic analysis of this device compared with historical data from the national database SNIIRAM will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a solid tumor.
2. Patient starting a first cycle of chemotherapy (+ - targeted therapy).
3. Patient starting intravenous chemotherapy including 21-day cycles.
4. Patient ≥18 years old.
5. Patient affiliated to a social security system in France.
6. Patient who signed the informed consent before study inclusion and before any study specific procedure.

Exclusion Criteria:

1. Patient already included in another interventional biomedical research.
2. Patient who began intravenous chemotherapy.
3. Patient who must receive an oral chemotherapy.
4. Patient who must be treated with a weekly chemotherapy or with concomitant radiotherapy.
5. Patient unreachable by phone.
6. Patient with no caregiver who can answer the phone in his place.
7. Pregnant or breastfeeding women.
8. Any psychological condition, family, geographic or social not to comply with medical monitoring and / or procedures in the study protocol.
9. Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Efficacy : Proportion of patients for which there was a modification in their care through the nurse device | 24 months

SECONDARY OUTCOMES:
Safety according to the classification of the CTCAE (Common for Toxicity Criteria for Adverse effects) V4.0 | 24 months
Quality of life using the QLQ-C30 questionnaire and the Skindex®-16 questionnaire | 24 months
Cost of the follow-up nursing device for the establishing | 24 months
Medical costs | 24 months
  Direct medical and non-medical costs of patients with malignant disease and followed by COACH will be compared to those of patients with the same types of cancer pathologies with traditional monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre DELORD, PhD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut claudius regaud, Toulouse, France